CLINICAL TRIAL: NCT01157429
Title: D-cycloserine Adjunctive Treatment for PTSD in Adolescents
Brief Title: D-cycloserine Adjunctive Treatment for Posttraumatic Stress Disorder (PTSD) in Adolescents
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Tulane University School of Medicine (Other)
Collaborators: National Alliance for Research on Schizophrenia and Depression (Other)
Responsible Party: Principal Investigator, Michael S. Scheeringa, Professor, Tulane University School of Medicine
Organization: Tulane University (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Tulane-09-00450
Record Dates: First submitted 2010-07-06; First posted 2010-07-07 (Estimated); Results first posted 2017-06-06 (Actual); Last update posted 2017-06-06 (Actual); Status verified 2017-04

CONDITIONS: Posttraumatic Stress Disorder; PTSD
Keywords: Cognitive Behavior Therapy; Children; Adolescents; Pharmacotherapy
MeSH Terms: conditions — Stress Disorders, Post-Traumatic | interventions — Cycloserine; Cognitive Behavioral Therapy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- D-cycloserine plus CBT (Active Comparator): Individuals receive 12 sessions of manualized trauma-focused cognitive behavioral therapy plus seven doses of D-cycloserine.
  Interventions: Drug: D-cycloserine; Behavioral: CBT
- Placebo pill (Placebo Comparator): Individuals receive 12 sessions of trauma-focused cognitive behavioral therapy plus seven doses of placebo pill.
  Interventions: Drug: Placebo pill; Behavioral: CBT

INTERVENTIONS:
Drug: D-cycloserine — D-cycloserine 50 mg by mouth prior to sessions 5-12 of the 12-session CBT protocol.
  Other Names: Seromycin
  Arms: D-cycloserine plus CBT
Drug: Placebo pill — Placebo pill by mouth prior to sessions 5-12 of teh 12-session CBT protocol.
  Arms: Placebo pill
Behavioral: CBT — 12-session CBT protocol, called Youth PTSD Treatment.
  Other Names: cognitive behavioral therapy

SUMMARY:
The purpose of this study is to show whether D-cycloserine in combination with cognitive behavioral therapy (CBT) is more effective than CBT plus placebo to reduce symptoms of posttraumatic stress disorder (PTSD) in 13-18 year-old children.

DETAILED DESCRIPTION:
While most individuals with PTSD treated with cognitive behavioral therapy (CBT) show improvement, they still have some enduring symptoms and functional impairment. Accordingly, there is a need for treatment advances. D-cycloserine (DCS), an antibiotic that has been used for over 50 years, has also been found to have positive effects on cognition and anxiety. DCS was found to enhance learning and memory, and also facilitates extinction of fear reactions. However, DCS only produces an extinction effect when paired with behavioral training, not when simply given alone. Thus, the medication only needs to be given for seven doses in this research and youth do not need to take the medication long term. The research also includes a three-month follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Certain number of PTSD symptoms plus functional impairment
* Must be able to swallow pills

Exclusion Criteria:

* Serious kidney or liver disease
* Epilepsy
* Bipolar disorder
* Psychosis

Ages: 13 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 24 (Actual)
Dates: Start 2010-06; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael S Scheeringa, MD, MPH, Principal Investigator — Tulane University School of Medicine
Locations (1):
- Tulane University Health Sciences Center, 1440 Canal St., New Orleans, Louisiana, United States

REFERENCES:
- [Derived] Scheeringa MS, Lilly ME, Staiger AB, Heller ML, Jones EG, Weems CF. Do Children and Adolescents Have Different Types of Trauma Narratives and Does It Matter? Reliability and Face Validation for a Narrative Taxonomy. J Trauma Stress. 2017 Jun;30(3):323-327. doi: 10.1002/jts.22190. Epub 2017 Jun 1. PMID 28569390
- [Derived] Scheeringa MS, Weems CF. Randomized placebo-controlled D-cycloserine with cognitive behavior therapy for pediatric posttraumatic stress. J Child Adolesc Psychopharmacol. 2014 Mar;24(2):69-77. doi: 10.1089/cap.2013.0106. Epub 2014 Feb 7. PMID 24506079

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 63 youth were assessed. Only 47 meet all the inclusion and exclusion criteria and were offered treatment. Of those 47, only 24 were retained through session 5 of the treatment, which was the point of random allocation. Twenty-three subjects of the 47 subjects who were offered treatment dropped out prior to session 5.
Groups:
- Placebo Pill: Individuals receive 12 sessions of trauma-focused cognitive behavioral therapy plus seven doses of placebo pill.
  Placebo pill: Placebo pill by mouth prior to sessions 5-12 of the 12-session CBT protocol.
Period: Overall Study
Arm/Group | D-cycloserine Plus CBT | Placebo Pill
Started | 12 | 12
Completed | 8 | 8
Not Completed | 4 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | D-cycloserine Plus CBT | Placebo Pill | Total
Number analyzed (Participants) | 12 | 12 | 24
Age, Continuous [Mean (Standard Deviation); unit: years] | 15.7 (1.6) | 15.9 (1.7) | 15.8 (1.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 7 | 17
  Male | 2 | 5 | 7
Region of Enrollment [Number; unit: participants]
  United States | 12 | 12 | 24

OUTCOME MEASURES:

1. Primary Outcome: Child PTSD Symptom Scale (CPSS)
Description: The CPSS is a 17-item standardized, self-administered questionnaires with versions for both youths and caregivers. Items are scored on 0-3 scale. Minimum possible score is 0 and maximum is 51. Only the total score is used; there are no subscales. A higher score indicates greater symptom severity (worse).
Time Frame: After 12 therapy sessions, up to 28 weeks.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | D-cycloserine Plus CBT | Placebo Pill
Number analyzed (Participants) | 8 | 8
units on a scale | 20.4 (9.7) | 11.0 (8.9)

ADVERSE EVENTS:
Time Frame: 2 months
Arm/Group | D-cycloserine Plus CBT | Placebo Pill
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/12
Other Adverse Events (participants affected / at risk) | 1/12 | 2/12
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | D-cycloserine Plus CBT (N=12) | Placebo Pill (N=12)
drowsy (Nervous system disorders) | 1 (2) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No